CLINICAL TRIAL: NCT01117987
Title: An Extension to QTI571A2301 to Evaluate the Long-term Safety, Tolerability and Efficacy of Oral QTI571 (Imatinib) in the Treatment of Severe Pulmonary Arterial Hypertension: IMPRES Extension
Brief Title: Extension to QTI571A2301 to Evaluate the Long-term Safety, Tolerability and Efficacy of Imatinib in Severe Pulmonary Arterial Hypertension (PAH)
Acronym: IMPRES Extn
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Novartis discontinued the development of imatinib in PAH due to requirement of regulatory authorities for additional data to secure marketing approval in PAH.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQTI571A2301E1; 2009-018167-26
Record Dates: First submitted 2010-05-03; First posted 2010-05-06 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension, imatinib, 6MWD, pulmonary hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Core imatinib (Experimental): Depending on the participants' randomized treatment in the core study, CQTI571A2301 (NCT00902174), and their completion status in the core study, participants received imatinib at 200 mg qd, 400 mg qd, or 200 mg qd with an increase to 400 mg qd after 2 weeks, if tolerated.
  Interventions: Drug: Imatinib; Drug: Placebo
- Core placebo (Experimental): Depending on the participants' randomized treatment in the core study, CQTI571A2301 (NCT00902174), and their completion status in the core study, participants received imatinib at 200 mg qd, 400 mg qd, or 200 mg qd with an increase to 400 mg qd after 2 weeks, if tolerated.
  Interventions: Drug: Imatinib; Drug: Placebo

INTERVENTIONS:
Drug: Imatinib — Participants, who received imatinib 200 mg in the core study, CQTI571A2301 (NCT00902174), and completed the core study, received imatinib 200 mg every day (qd) in the extension. Participants, who were randomized to receive imatinib 400 mg in the core study and completed the core study, received imatinib 400 mg qd in the extension. Participants, who terminated early from the core study or who were randomized to placebo and completed the core study, started the extension with imatinib 200 mg qd. After 2 weeks, the dose was increased to 400 mg qd if tolerated.
Drug: Placebo — To preserve the blind of the core study until the core study, CQTI571A2301 (NCT00902174), was completed, participants received a blinded study drug package containing a 70-tablet bottle of imatinib and a 70-tablet bottle of matching placebo.

SUMMARY:
This is a multinational, multi center extension study. This study will provide data on the long-term safety, tolerability, and efficacy of imatinib in the treatment of severe pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who participated in CQTI571A2301 clinical trial and completed the week 24 visit of the study protocol, including all Study Completion assessments
* Patients who withdrew from the CQTI571A2301 study prematurely for reasons not related to study drug or not related to a safety issue but performed all Study Completion assessments

Exclusion Criteria:

* Patients with a pulmonary capillary wedge pressure > 15 mmHg at time of Study Completion assessments in core protocol CQTI571A2301. If pulmonary capillary wedge pressure is not attainable, then a left atrial pressure measurement may be used in its place.
* LVEF < 45%
* Patients with thrombocytopenia, platelet count < 50E9/L (50E3/µL)
* Patients with uncontrolled systemic arterial hypertension, systolic > 160 mmHg or diastolic > 90 mmHg
* Patients with a QTcF > 450 ms for males and > 470 ms for females in the absence of right branch bundle block (based on Visit 1 ECG if required to be performed)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (55):
- United States (19):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Weston, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tualatin, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Milwaulkee, Wisconsin
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Leuven, Belgium
- Canada (3):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, London, Ontario
- Novartis Investigative Site, Clamart, France
- Germany (11):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Würzburg
- Italy (2):
  - Novartis Investigative Site, Pavia, (pv)
  - Novartis Investigative Site, Roma, RM
- Japan (5):
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (5):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
- Novartis Investigative Site, Sankt Gallen, Switzerland
- United Kingdom (4):
  - Novartis Investigative Site, Cambridge, Cambridgeshire
  - Novartis Investigative Site, Newcastle upon Tyne, Newcastle
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, London

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Imatinib; Core Placebo: Depending on the participants randomized treatment in the core study, CQTI571A2301 (NCT00902174), and their completion status in the core study, participants received imatinib at 200 mg qd, 400 mg qd, or 200 mg qd with an increase to 400 mg qd after 2 weeks, if tolerated.
Period: Overall Study
Arm/Group | Core Imatinib | Core Placebo
Started | 66 | 78
Completed | 5 | 4
Not Completed | 61 | 74
Not completed — Protocol deviation | 0 | 1
Not completed — Subject no longer requires study drug | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Abnormal test procedure result | 2 | 0
Not completed — Lack of Efficacy | 3 | 4
Not completed — Death | 5 | 10
Not completed — Withdrawal by Subject | 5 | 10
Not completed — Adverse Event | 19 | 26
Not completed — Administrative problems | 25 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Imatinib | Core Placebo | Total
Number analyzed (Participants) | 66 | 78 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (15.52) | 45.7 (13.31) | 47.4 (14.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 63 | 120
  Male | 9 | 15 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Deaths
Description: Adverse event monitoring was conducted throughout the study.
Time Frame: 204 weeks
Population: Safety analysis set: The safety set included all paticipants who received at least one dose of study drug during the extension.
Measure: Number; unit: Participants
Arm/Group | Core Imatinib | Core Placebo
Number analyzed (Participants) | 66 | 78
Participants
  Adverse events (non-serious and serious) | 62 | 76
  Serious adverse events | 40 | 53
  Deaths | 6 | 10

2. Secondary Outcome: Change From Core Study Baseline in Six-Minute Walk Distance (6MWD)
Description: A six minute walk test (6MWT) was performed in accordance with the guidleines of the American Thoracic Society (2002).
Time Frame: core study baseline, extension baseline, 12 weeks, 24 weeks, 48 weeks, 72 weeks, 96 weeks, 120 weeks, 144 weeks, 156 weeks, 204 weeks
Population: Participants from the Full Analysis Set (FAS), who had values at both core study baseline and the given post-baseline time point, were included in the analysis for that post-baseline time point. The FAS included all participants who received at least one dose of study drug during the extension.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Core Imatinib | Core Placebo
Number analyzed (Participants) | 66 | 78
meters
  Extension baseline (n=61,77) | 42.98 (55.209) | 4.91 (62.629)
  Week 12 (n=58,57) | 48.75 (60.887) | 16.25 (64.992)
  Week 24 (n=54,53) | 44.71 (45.506) | 19.34 (71.675)
  Week 48 (n=47,42) | 45.81 (72.150) | 29.18 (65.198)
  Week 72 (n=40,39) | 49.54 (76.019) | 56.46 (111.130)
  Week 96 (n=38,35) | 66.64 (71.080) | 41.03 (54.495)
  Week 120 (n=32,29) | 83.19 (67.855) | 37.43 (60.087)
  Week 144 (n=27,21) | 67.70 (64.000) | 39.45 (79.356)
  Week 156 (n=21,18) | 72.60 (67.972) | 30.17 (66.856)
  Week 204 (n=4,3) | 96.88 (42.048) | 4.50 (25.608)

3. Secondary Outcome: Percentage of Participants With Incidence of Clinical Worsening Events
Description: Clinical worsening events included death, overnight hospitalization for worsening of PAH, worsening of World Health Organization (WHO) functional class by at least one level (drop in WHO ), 15% decrease in the 6MWD as compared to baseline confirmed by two 6MWTs at two consecutive study visits (6MWD reduction), and drop in WHO & 6MWD reduction. Some participants have fulfilled more than one criterion. Therefore, the sum of individual components may be higher than the total number of participants with clinical worsening.
Time Frame: 204 weeks
Population: Full Analysis Set (FAS): The full analysis set included all participants who received at least one dose of study drug during the extension.
Measure: Number; unit: Percentage of participants
Arm/Group | Core Imatinib | Core Placebo
Number analyzed (Participants) | 66 | 78
Percentage of participants
  Total participants with clinical worsening | 50.0 | 46.2
  Death (all deaths) | 7.6 | 12.8
  Hospitalization for worsening of PAH | 33.3 | 28.2
  Drop in WHO | 24.2 | 19.2
  6MWD reduction | 12.1 | 19.2
  Drop in WHO and 6MWD reduction | 1.5 | 3.8

ADVERSE EVENTS:
Arm/Group | Core Imatinib | Core Placebo
Serious Adverse Events (participants affected / at risk) | 40/66 | 53/78
Other Adverse Events (participants affected / at risk) | 55/66 | 72/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Imatinib (N=66) | Core Placebo (N=78)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Coagulopathy (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2
Cor pulmonale (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 5 | 8
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 1
Astigmatism (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Corneal erosion (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Brain death (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Device dislocation (General disorders) | 0 | 1
Device leakage (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 1
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 5 | 3
Device related sepsis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 3
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted lung (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Eosinophil percentage increased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0
N-terminal prohormone brain natriuretic peptide (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 2
Syncope (Nervous system disorders) | 2 | 7
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Scleroedema (Skin and subcutaneous tissue disorders) | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1
Craniotomy (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Imatinib (N=66) | Core Placebo (N=78)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 7
Palpitations (Cardiac disorders) | 4 | 4
Pericardial effusion (Cardiac disorders) | 0 | 4
Tachycardia (Cardiac disorders) | 4 | 4
Conjunctival haemorrhage (Eye disorders) | 2 | 5
Periorbital oedema (Eye disorders) | 11 | 23
Abdominal discomfort (Gastrointestinal disorders) | 2 | 5
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 18 | 27
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Gastritis (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 21 | 39
Vomiting (Gastrointestinal disorders) | 14 | 25
Asthenia (General disorders) | 4 | 2
Chest discomfort (General disorders) | 2 | 4
Face oedema (General disorders) | 1 | 4
Fatigue (General disorders) | 9 | 11
Non-cardiac chest pain (General disorders) | 4 | 4
Oedema peripheral (General disorders) | 21 | 32
Pyrexia (General disorders) | 9 | 5
Seasonal allergy (Immune system disorders) | 3 | 4
Bronchitis (Infections and infestations) | 1 | 8
Device related infection (Infections and infestations) | 0 | 4
Influenza (Infections and infestations) | 5 | 2
Nasopharyngitis (Infections and infestations) | 17 | 24
Pneumonia (Infections and infestations) | 1 | 4
Respiratory tract infection (Infections and infestations) | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 11
Urinary tract infection (Infections and infestations) | 3 | 8
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 4
Blood creatinine increased (Investigations) | 4 | 3
Weight decreased (Investigations) | 5 | 3
Weight increased (Investigations) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4
Fluid overload (Metabolism and nutrition disorders) | 1 | 4
Gout (Metabolism and nutrition disorders) | 2 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 10
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 5
Dizziness (Nervous system disorders) | 9 | 5
Headache (Nervous system disorders) | 12 | 24
Insomnia (Psychiatric disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 13
Flushing (Vascular disorders) | 2 | 5
Hypotension (Vascular disorders) | 6 | 3

LIMITATIONS AND CAVEATS:
Within primary outcome measure (OM) #1, an additional death (>30 days post study completion) was included in the imatinib arm. The participant flow and secondary OM #2 reflect deaths that occurred up to and including 30 days post study completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.